CLINICAL TRIAL: NCT00385073
Title: Assessing the Role of Exercise Intensity in Slowing Disease Progression in Early Parkinson's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Austin Health (Other Government)
Other Study IDs: 126/05
Record Dates: First submitted 2006-10-05; First posted 2006-10-06 (Estimated); Last update posted 2006-10-06 (Estimated); Status verified 2006-10

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Participants will complete a self-selected intensity of exercising over a 6 month period, with detailed clinical assessments at commencement and completion to determine the rate of progression of parkinsonism and gait abnormalities

DETAILED DESCRIPTION:
Participants will complete a self-selected intensity of exercising over a 6 month period - including jogging, swimming and circuit training, with detailed clinical assessments at commencement and completion (including UPDRS, gaitrite lab study) to determine the rate of progression of parkinsonism and gait abnormalities

ELIGIBILITY:
Inclusion Criteria:

* Early Parkinson's Disease,
* Able to provide informed consent,
* able to complete exercise diaries for 6 months,
* no medications or on levo-dopa

Exclusion Criteria:

* Not on dopamine agonists,

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2005-04; Study Completion 2007-12

CONTACTS AND LOCATIONS:
Overall Officials: mary m galea, PgD, Principal Investigator — Austin Health
Locations (1):
- Royal Talbot Rehabilitation Centre, Melbourne, Australia